CLINICAL TRIAL: NCT03886701
Title: A Phase 1, Open-Label, Fixed-Sequence, Drug Interaction Study to Investigate the Effect of Once-Weekly Rifapentine and Isoniazid on the Pharmacokinetics of Steady-State Doravirine
Brief Title: Doravirine, Rifapentine and Isoniazid Interaction
Acronym: DORIIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Walter K. Kraft (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Walter K. Kraft, Principal Investigator, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12690
Record Dates: First submitted 2019-03-12; First posted 2019-03-22 (Actual); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Latent Tuberculosis; Human Immunodeficiency Virus; Rifamycins Causing Adverse Effects in Therapeutic Use; Drug Interaction Potentiation
Keywords: Drug-drug interaction; Pharmacokinetics; Non-nucleoside reverse transcriptase inhibitor; NNRTI; LTBI; Antimycobacterial
MeSH Terms: conditions — Latent Tuberculosis; Acquired Immunodeficiency Syndrome | interventions — doravirine; rifapentine; Isoniazid; Drugs, Generic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Period 1: DOR twice-daily alone (Study days 1-4) and Period 2: DOR twice-daily with RPT and INH once-weekly (Study days 7-21)
  Interventions: Drug: Doravirine (DOR); Drug: Rifapentine (RPT); Drug: Isoniazid (INH)

INTERVENTIONS:
Drug: Doravirine (DOR) — Non-nucleoside reverse transcriptase inhibitor indicated for the treatment of HIV-1 infection in adults in combination with other antiretroviral agents.
  Other Names: Pifeltro
Drug: Rifapentine (RPT) — Rifamycin anti-tuberculosis agent indicated for the treatment of latent and active tuberculosis infection.
  Other Names: Priftin
Drug: Isoniazid (INH) — Anti-tuberculosis agent indicated for the treatment of latent and active tuberculosis infection.
  Other Names: Generic (various)

SUMMARY:
Drug therapy for persons living with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) co-infected with latent tuberculosis infection (LTBI) is complex. Anti-tuberculosis drugs used to treat LTBI often induce drug metabolizing enzymes that share the same metabolic pathway as antiretroviral drugs used for those living with HIV/AIDS. This study evaluates the drug-drug interaction (DDI) potential of an antiretroviral drug when co-administered with a common anti-tuberculosis regimen of drugs.

DETAILED DESCRIPTION:
Rifapentine (RPT) and isoniazid (INH) given once weekly for 12 weeks is commonly used for treating LTBI in adults. For people living with HIV-1, the risks of LTBI is increased. Individuals living with HIV-1 are often on chronic antiretroviral drugs that prevent immunodeficiency and complications associated with infection. Unfortunately, antiretroviral drugs are subject to many DDIs especially with RPT which induces drug clearing enzymes.

Doravirine (DOR) is a newly approved non-nucleoside reverse transcriptase inhibitor indicated for the treatment of HIV-1 infection. Because RPT induces the metabolic pathway in which DOR is removed, there is concern that taking both concomitantly will result in an unwanted DDI leading to reduced DOR concentrations in the blood. Reduced levels will result in loss of efficacy for the drug and therefore not provide adequate viral suppression in those living with HIV. This study investigates the DDI potential of the once weekly regimen RPT and INH together with DOR in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between 18-60 years old at the time of screening.
2. Have a Body Mass Index (BMI) > 19 and < 33.
3. Weigh > 45 kg but < 120 kg.
4. Non-smoker (tobacco or electronic cigarettes).
5. Negative QuantiFERON-TB Gold at screening.
6. Subjects who agree to abstain from alcohol consumption throughout the duration of the study.
7. Female subjects of childbearing potential must demonstrate a urine beta-hCG consistent with non-pregnancy at the time of the screening visit and agree to the use (and/or have their partner use) of an acceptable method of birth-control at initial screening, during the time of the trial and until two weeks after the last dose of drug following the last treatment period.
8. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, dermatologic, psychiatric abnormalities or neurological (including stroke and chronic seizure) diseases.
2. >500 mL blood or plasma donation in the 6 weeks prior to study start
3. Known anaphylactic or severe systemic reactions to any components of doravirine, rifapentine, isoniazid or pyridoxine.
4. Positive HIV, Hepatitis B or Hepatitis C virus. Evidence of prior Hepatitis B infection and immunity is not exclusionary.
5. Latent or active tuberculosis infection. Documented prior fully treated latent tuberculosis is not exclusionary.
6. Females who are postpartum < 12 months.
7. Current drug or alcohol abuse.
8. Received study drug in another study within 4 weeks or within 5 half-lives, which ever occurring first, before first anticipated dose of study drug in this study.
9. Unable to refrain from use of over-the-counter, prescription (unless determined appropriate by the investigator), herbal or natural products, vitamins or supplements, or grapefruit juice/grapefruit products.
10. Any clinical significant findings on lab, ECG or physical exam at screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter K Kraft, MD, Principal Investigator — Sidney Kimmel Medical College at Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Clinical Research Unit, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Particpants: Eleven healthy volunteers enrolled into the study. For period 1 (study days 1-4), participants will be given doravirine 100mg oral tablets dosed twice-daily on study days 1-4. For period 2 (study days 7-21), oral 100mg doravirine will be dosed twice-daily. Weight-based rifapentine and isoniazid (as recommended by the CDC) will be given orally once-weekly on study days 7, 14, and 21.
Period: Period 1: Study Days 1-4
Arm/Group | Study Particpants
Started (Healthy volunteers received oral DOR 100 mg twice daily alone) | 11
Completed | 11
Not Completed | 0
Period: Period 2: Study Days 7-21
Arm/Group | Study Particpants
Started (Healthy volunteers received oral DOR 100 mg twice daily together with once weekly RPT and INH) | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Particpants: Eleven healthy volunteers enrolled into the study.
Arm/Group | Study Particpants
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 50 [27 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3
  Black or African American | 8
Weight [Mean (Standard Deviation); unit: Kilogram] | 92.9 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Doravirine Maximum Concentration (Cmax)
Description: Doravirine maximum observed concentration during the dosing interval
Time Frame: Day 4 and 21 (Period 1 and 2): 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Groups:
- Period 1: DOR twice-daily alone (Study days 1-4)
  Doravirine (DOR): Non-nucleoside reverse transcriptase inhibitor indicated for the treatment of HIV-1 infection in adults in combination with other antiretroviral agents.
  Rifapentine (RPT): Rifamycin anti-tuberculosis agent indicated for the treatment of latent and active tuberculosis infection.
  Isoniazid (INH): Anti-tuberculosis agent indicated for the treatment of latent and active tuberculosis infection.
- Period 2: DOR twice-daily with RPT/INH once-weekly (Study days 7-21)
Arm/Group | Period 1 | Period 2
Number analyzed (Participants) | 11 | 11
ug/mL | 1.7 [1.5 to 2] | 1.3 [1.1 to 1.5]

2. Primary Outcome: Doravirine Area Under the Plasma Concentration Versus Time Curve From 0 to 12 Hours (AUC0-12)
Description: Doravirine area under the plasma-concentration time curve derived from plasma sampling during one dosing interval
Time Frame: Day 4 and 21 (Period 1 and 2): 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Measure: Geometric Mean (95% Confidence Interval); unit: hr x ug/mL
Arm/Group | Period 1 | Period 2
Number analyzed (Participants) | 11 | 11
hr x ug/mL | 17.3 [14.9 to 20] | 12.3 [10.4 to 14.3]

3. Primary Outcome: Doravirine Oral Clearance (CL/F)
Description: Doravirine apparent oral clearance derived from plasma sampling
Time Frame: Day 4 and 21 (Period 1 and 2): 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Period 1 | Period 2
Number analyzed (Participants) | 11 | 11
L/hr | 5.9 (24) | 8.4 (26.1)

4. Secondary Outcome: Adverse Event
Description: Safety and tolerability
Time Frame: Days 1-24 post-dose (period 1 and 2) and 31-34 post-dose (post-study)
Measure: Number; unit: participants
Arm/Group | Period 1 | Period 2
Number analyzed (Participants) | 11 | 11
participants
  Nausea/vomiting | 1 | 0
  Dysuria | 0 | 1
  Fever | 0 | 1
  Headache | 0 | 1
  Chills | 0 | 1
  Catheter site pain and redness | 3 | 2

ADVERSE EVENTS:
Time Frame: Daily for the duration of the study and 7-10 days post-study.
Arm/Group | Period 1 | Period 2
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 4/11 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1 (N=11) | Period 2 (N=11)
Nausea/vomiting (Gastrointestinal disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Catheter site pain and redness (General disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03886701/Prot_SAP_000.pdf